CLINICAL TRIAL: NCT02894112
Title: Effects of Fluid Milk in Attenuating Hyperglycemia and Hypertriglyceridemia After Meal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Dairy Research Institute (Other)
Responsible Party: Principal Investigator, Miriam Pearman-Leary, Doctoral Candidate, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1198
Record Dates: First submitted 2016-08-30; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Oral Glucose Tolerance Test; High Fat Tolerance Test
Keywords: endothelial dependent vasodilation; blood flow; blood glucose; triglycerides; non-fat milk; dairy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral glucose tolerance test (Experimental): 100 g of glucose in a fruit punch flavored 8 oz drink
  Interventions: Dietary Supplement: non-fat milk; Dietary Supplement: carbohydrate control beverage; Dietary Supplement: caloric control beverage
- High fat tolerance test (Experimental): single high fat load determined by body weight.
  Interventions: Dietary Supplement: non-fat milk; Dietary Supplement: carbohydrate control beverage; Dietary Supplement: caloric control beverage

INTERVENTIONS:
Dietary Supplement: non-fat milk — 1 serving of non-fat fluid milk
Dietary Supplement: carbohydrate control beverage — 1 serving of carbohydrate control beverage (Carbohydrate powder + water)
Dietary Supplement: caloric control beverage — 1 serving of caloric control beverage (carbohydrate powder + protein powder + water)

SUMMARY:
Epidemiological studies indicate that risk of type 2 diabetes is lower when milk is consumed in the regular diet. Milk products are unique in that they produce high insulin response despite their low glycemic index. The general aim of the proposed study is to determine the effect of fluid milk on attenuating the postprandial surge in plasma glucose and triglyceride after meals and its associated physiological mechanisms. The investigators hypothesize that the consumption of one or two servings of non-fat milk added to a standard oral glucose tolerance test (OGTT) solution or the high fat tolerance test meal will attenuate postprandial hyperglycemia and triglyceridemia. The investigators hypothesize that the postulated improvement in postprandial metabolic response due to the consumption of fluid milk will be associated with increased postprandial insulin secretion as well as insulin-mediated endothelial vasodilation and whole-limb perfusion.

DETAILED DESCRIPTION:
A double blind randomized placebo-controlled crossover experimental design with six treatments will be used. A total of 30 young (20-40 year old) healthy men and women will serve as subjects. Following 2 days of physical activity and dietary control, subjects will consume a standard OGTT load or high fat tolerance load on the morning of Day 3. The solution used in the meals will be mixed with one or two servings of non-fat milk or placebo (either carbohydrate matched or total calorie matched). Before and after the test meals are consumed, blood samples will be obtained for later analysis of glucose, triglycerides, insulin, and inflammatory cytokines and brachial artery flow-mediated dilation and femoral artery vascular conductance will be measured. The present research project should provide new and clinically useful insight into the role of conventional dairy products on metabolic homeostasis. If the working hypotheses are supported, the information could be used as an initial/preliminary basis for recommendations for the consumption of fluid milk in the prevention of metabolic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Apparently health, sedentary. All subjects will have a BMI of 25-35 kg/m2.

Exclusion Criteria:

* Candidates who are taking cardiovascular-acting drugs will not be eligible for participation. Subjects with significant intima-media thickening, plaque formation, characteristics of atherosclerosis, metabolic diseases, gastrointestinal disorders, and/or renal disease will be excluded from the study. Additional exclusion criteria will be cow milk allergy or lactose intolerance, pregnancy or lactation, and alcohol abuse.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
blood glucose | 2 hour postprandially
plasma triglyceride | 4 hour postprandially

SECONDARY OUTCOMES:
femoral artery blood flow | 2-4 hour postprandially
brachial artery flow-mediated dilation | 2-4 hour postprandially

OTHER OUTCOMES:
insulin | 2-4 hour postprandially
glucagon | 2-4 hour postprandially
GIP | 2-4 hour postprandially
GLP | 2-4 hour postprandially

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Aging Research Laboratory, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No